CLINICAL TRIAL: NCT04844385
Title: A Prospective Single-arm Phase Ⅱ Study of Toripalimab Plus Neoadjuvant Chemotherapy Combined With Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma
Brief Title: Toripalimab Plus Neoadjuvant Chemotherapy Combined With Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1071
Record Dates: First submitted 2021-03-01; First posted 2021-04-14 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Toripalimab, Neoadjuvant, Concurrent Chemoradiotherapy, Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; nedaplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients in cohort A receive 2 cycles Toripalimab plus Paclitaxel/Nedaplatin, followed by radiotherapy at a total dose of 60Gy combined with Capecitabine.
  Interventions: Drug: Toripalimab; Drug: Paclitaxel-albumin; Drug: Nedaplatin; Radiation: radiation therapy at a total dose 60 Gy; Drug: Capecitabine
- Cohort B (Experimental): Patients in cohort B receive 2 cycles Toripalimab plus Paclitaxel/Nedaplatin, followed by radiotherapy at a total dose of 50Gy combined with Capecitabine.
  Interventions: Drug: Toripalimab; Drug: Paclitaxel-albumin; Drug: Nedaplatin; Drug: Capecitabine; Radiation: radiation therapy at a total dose 50 Gy

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240 mg, d1, Q3w for two cycles
Drug: Paclitaxel-albumin — Paclitaxel-albumin 260 mg/m2, d1, Q3w for two cycles
Drug: Nedaplatin — Nedaplatin 75mg/m2, d1, Q3w for two cycles
Radiation: radiation therapy at a total dose 60 Gy — Radiation therapy at a total dose 60 Gy
  Arms: Cohort A
Drug: Capecitabine — Capecitabine 1000 mg/m2, bid, d1-14, q3w during radiotherapy
Radiation: radiation therapy at a total dose 50 Gy — Radiation therapy at a total dose 50 Gy
  Arms: Cohort B

SUMMARY:
This Phase II non-randomized study is to determine the efficacy and toxicity of neoadjuvant toripalimab plus chemotherapy followed by chemoradiotherapy for locally advanced unresectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This Phase II non-randomized study is to determine the efficacy and toxicity of neoadjuvant toripalimab plus chemotherapy followed by chemoradiotherapy for locally advanced unresectable esophageal squamous cell carcinoma.

All patients were planned to receive 2 cycle of toripalimab plus paclitaxel/nedaplatin as neoadjuvant therapy. Then they all receive radical dose of chest radiation and concurrent chemotherapy of capecitabine (PO 1000 mg/m2, bid, d1-d14, q3w).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed esophageal squamous cell carcinoma
* patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* unresectable T1-4 N0-3 M0-1 confirmed by CT or MRI (M1 only includes patients with lymph node metastasis in the supraclavicular region)
* ECOG performance status 0-1
* no previous chest radiotherapy, immunotherapy or biotherapy.
* hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ
* contraindication for chemotherapy
* women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* women who has the probability of pregnancy without contraception
* tendency of hemorrhage
* in other clinical trials within 30 days
* addicted in drugs or alcohol, AIDS patients
* uncontrollable seizure or psychotic patients without self-control ability
* severe allergy or idiosyncrasy
* not suitable for this study judged by researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate | 18-month

SECONDARY OUTCOMES:
overall survival rate | 18-month
Clinical response rate | 2 months after radiotherapy
  the percentage of patients who had partial remission or complete remission after therapy
the rate of grade 3 or 4 toxicities according to CTCAE4.0 | 1 year after therapy
  the percentage of patients who develop grade 3 or 4 toxicities
distant metastasis-free survival | 18-month
locoregional recurrence-free survival | 18-month
Quality of life assessed by QLQ-C30 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Background] Gaspar LE, Winter K, Kocha WI, Coia LR, Herskovic A, Graham M. A phase I/II study of external beam radiation, brachytherapy, and concurrent chemotherapy for patients with localized carcinoma of the esophagus (Radiation Therapy Oncology Group Study 9207): final report. Cancer. 2000 Mar 1;88(5):988-95. PMID 10699886
- [Background] Kojima T, Shah MA, Muro K, Francois E, Adenis A, Hsu CH, Doi T, Moriwaki T, Kim SB, Lee SH, Bennouna J, Kato K, Shen L, Enzinger P, Qin SK, Ferreira P, Chen J, Girotto G, de la Fouchardiere C, Senellart H, Al-Rajabi R, Lordick F, Wang R, Suryawanshi S, Bhagia P, Kang SP, Metges JP; KEYNOTE-181 Investigators. Randomized Phase III KEYNOTE-181 Study of Pembrolizumab Versus Chemotherapy in Advanced Esophageal Cancer. J Clin Oncol. 2020 Dec 10;38(35):4138-4148. doi: 10.1200/JCO.20.01888. Epub 2020 Oct 7. PMID 33026938
- [Background] Kato K, Shah MA, Enzinger P, Bennouna J, Shen L, Adenis A, Sun JM, Cho BC, Ozguroglu M, Kojima T, Kostorov V, Hierro C, Zhu Y, McLean LA, Shah S, Doi T. KEYNOTE-590: Phase III study of first-line chemotherapy with or without pembrolizumab for advanced esophageal cancer. Future Oncol. 2019 Apr;15(10):1057-1066. doi: 10.2217/fon-2018-0609. Epub 2019 Feb 8. PMID 30735435
- [Background] Fan TY, Xing J, Lu J, Liu TH, Xu M, Zhang YJ, Shao Q, Li JB, Yu JM. Phase I/II study of induction chemotherapy plus concurrent chemotherapy and SMART-IMRT-based radiotherapy in locoregionally-advanced nasopharyngeal cancer. Oncol Lett. 2013 Mar;5(3):889-895. doi: 10.3892/ol.2013.1137. Epub 2013 Jan 15. PMID 23426016
- [Background] Koom WS, Kim TH, Shin KH, Pyo HR, Kim JY, Kim DY, Yoon M, Park SY, Lee DH, Ryu JS, Jung YS, Lee SH, Cho KH. SMART (simultaneous modulated accelerated radiotherapy) for locally advanced nasopharyngeal carcinomas. Head Neck. 2008 Feb;30(2):159-69. doi: 10.1002/hed.20667. PMID 17764088
- [Background] Butler EB, Teh BS, Grant WH 3rd, Uhl BM, Kuppersmith RB, Chiu JK, Donovan DT, Woo SY. Smart (simultaneous modulated accelerated radiation therapy) boost: a new accelerated fractionation schedule for the treatment of head and neck cancer with intensity modulated radiotherapy. Int J Radiat Oncol Biol Phys. 1999 Aug 1;45(1):21-32. doi: 10.1016/s0360-3016(99)00101-7. PMID 10477002
- [Background] Welsh J, Palmer MB, Ajani JA, Liao Z, Swisher SG, Hofstetter WL, Allen PK, Settle SH, Gomez D, Likhacheva A, Cox JD, Komaki R. Esophageal cancer dose escalation using a simultaneous integrated boost technique. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):468-74. doi: 10.1016/j.ijrobp.2010.10.023. Epub 2010 Dec 1. PMID 21123005
- [Background] Song YP, Ma JB, Hu LK, Zhou W, Chen EC, Zhang W. Phase I/II study of hypofractioned radiation with three-dimensional conformal radiotherapy for clinical T3-4N0-1M0 stage esophageal carcinoma. Technol Cancer Res Treat. 2011 Feb;10(1):25-30. doi: 10.7785/tcrt.2012.500176. PMID 21214285
- [Background] Ma JB, Wei L, Chen EC, Qin G, Song YP, Chen XM, Hao CG. Moderately hypofractionated conformal radiation treatment of thoracic esophageal carcinoma. Asian Pac J Cancer Prev. 2012;13(8):4163-7. doi: 10.7314/apjcp.2012.13.8.4163. PMID 23098423
- [Derived] Liu F, Wang D, Rong Y, Wei S, SiTu Y, Wang M, Zhang H, Zhang P, Zheng S, Yin S, Xie C, Hu Y, Qiu B, Liu H. Safety and efficacy of neoadjuvant toripalimab plus chemotherapy followed by chemoradiotherapy for locally advanced esophageal squamous cell carcinoma in China (GASTO 1071): a non-randomised, two-cohort, phase 2 trial. EClinicalMedicine. 2025 Apr 5;82:103184. doi: 10.1016/j.eclinm.2025.103184. eCollection 2025 Apr. PMID 40242562